CLINICAL TRIAL: NCT06612515
Title: Prospective Cohort-study for the Investigation of the Vac-cine-induced Immune Response After Vaccination Against RESPiratory Viral Infections in Immunocompromised Pa-tients With or Without Haemato-ONcological diseaSEs
Brief Title: Vaccine-induced Immunity in Immunocompromised Patients
Acronym: RESPONSE
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Sibylle C Mellinghoff, Board certified medical doctor, University of Cologne
Other Study IDs: 231244-NIS
Record Dates: First submitted 2024-09-19; First posted 2024-09-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Immunodeficiency
Keywords: vaccine; Immunocompromised; immune response
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA and Serum blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Managing respiratory virus infections in immunocompromised patients requires a multidisciplinary approach, including vaccination, though its effectiveness is often suboptimal in these individuals.

In hematological patients, poor humoral immunogenicity is common, especially when the B cell axis is affected by disease or treatment, while T cell responses may offer better protection. Current immunologic data on these patients is limited, focusing mostly on serologic parameters. To address this, we will conduct an observational study analyzing early and late booster vaccinations, with a focus on virus-specific T cell responses in vaccinated patients.

DETAILED DESCRIPTION:
Respiratory virus infections are a significant cause of morbidity and mortality, partic-ularly among immunocompromised patients. These infections are caused by a varie-ty of viral pathogens, including influenza viruses, respiratory syncytial virus (RSV), parainfluenza viruses, adenoviruses, rhinoviruses, and coronaviruses, among oth-ers. In the general population, these infections typically result in self-limiting ill-nesses; however, in individuals with compromised immune systems, such as those undergoing chemotherapy, organ transplant recipients, patients with haematological malignancies, and those with HIV, the consequences can be severe and often life-threatening. For example, patients with haematological and oncological diseases are at elevated risk for severe morbidity and mortality by influenza infections. Com-pared to influenza-associated hospitalization rates in the general population (37.9 per 100,000 person-years for persons age 50 to 64 years)1 patients with cancer were hospitalized at a rate of 219 per 100,000 person-years for patients younger than 65 years.

The immune system plays a crucial role in defending against viral pathogens. Im-munocompromised patients, due to either primary immune deficiencies or second-ary immunosuppression (e.g., from immunosuppressive therapies), have impaired immune responses that hinder the effective clearance of viral infections. This im-pairment can lead to prolonged viral shedding, increased risk of secondary bacterial infections, and more severe disease manifestations, including acute respiratory dis-tress syndrome (ARDS) and multi-organ failure. The management of respiratory vi-rus infections in immunocompromised patients requires a multidisciplinary ap-proach. Prophylactic measures, including vaccination and the use of antiviral prophylaxis, are crucial in reducing the incidence of these infections.

Given the significant impact of respiratory virus infections on immunocompromised patients, ongoing research is crucial to improve preventive strategies. This research includes studies on viral pathophysiology, host immune responses, and the devel-opment of optimal vaccination schedules. The emergence of new viral pathogens, such as SARS-CoV-2, underscores the importance of surveillance and prepared-ness in this vulnerable population.

Respiratory virus infections represent a major health concern for immunocompro-mised patients, necessitating comprehensive and specialised care. Continued ad-vancements in diagnostics, therapeutics, and preventive measures are vital to miti-gate the impact of these infections and improve the quality of life and survival of immunocompromised individuals.

The management of respiratory virus infections in immunocompromised patients requires a multidisciplinary approach and prophylactic measures, including vaccina-tion, to reduce the incidence and severity of these infections. However, the efficacy of vaccination is often suboptimal in immunocompromised individuals and not well assessed in clinical trials.

A poor humoral immunogenicity has been shown for most available vaccines in haematological patients. Especially affection of the B cell axis by either disease, treatment, or both, impacts humoral vaccine immune response.

The humoral vaccine-induced immune response facilitates early protection directly after vaccination, while long-term protection warrants antibody persistence as well as immune memory cells. Data from immunocompetent persons suggest that cell mediated immune response may be a better correlate of protection against virus in-fections in vaccinated patients with poor immune responses than humoral im-munity due to its major role in recovery from infection and in virus clearance.

Immunologic data in patients with haematological malignancies are generally scarce and mainly focus on serologic parameters. However, cellular response and especially T cell response seems often to be induced more reliably in those patients than humoral response as seen in other immunocompromised populations18 and other vaccines.

To close this knowledge gap, we will perform an observational study to prospectively analyse the effect of early and late booster vaccination with special focus on the virus-specific T cells. Samples will be collected from patients that have been vac-cinated as part of clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Patients with immunosuppression either by treatment or underlying diseases
* Patients who are vaccinated or willing to be vaccinated against respiratory virus infections in ac-cordance with current recommendations
* Age of 18 years or older

Exclusion Criteria:

* Patients unwilling/ineligible for vaccination under current recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Immunocompromised patients vaccinated against respiratory virus infections or willing to be vaccinated
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response after vaccination | 12 months
  To compare antibody titres between different subgroups of immunocompromised patients after vaccination against respiratory virus infections

SECONDARY OUTCOMES:
Cellular immune response after vaccination | 12 months
  To analyse T cell response after vaccination against respiratory virus infections
Seroconversion | 12 months
  To compare antibody response rates between dif-ferent subgroups of immunocompromised patients after vaccination against respiratory virus infections

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany